CLINICAL TRIAL: NCT05624060
Title: The Effect of Perineal Massage and Pelvic Floor Exercise Applied in the Antenatal Period on Postpartum Sexuality and Incontinence: a Randomized Controlled Study
Brief Title: Perineal Massage and Pelvic Floor Exercise in the Antenatal Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan OZKAN SAT, Assistant Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SULTANOZKANSAT
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-11

CONDITIONS: Urinary Incontinence; Fecal Incontinence; Sexual Dysfunction; Sexuality
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence; Sexual Dysfunction, Physiological; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): Pelvic Floor Dysfunction Prevention Training
  Interventions: Behavioral: Pelvic Floor Dysfunction Prevention Training
- Experimental Group 1 (Experimental): Pelvic Floor Dysfunction Prevention Training and Perineal Massage
  Interventions: Behavioral: Pelvic Floor Dysfunction Prevention Training; Behavioral: Pelvic Floor Dysfunction Prevention Training and Perineal Massage
- Experimental Group 2 (Experimental): Pelvic Floor Dysfunction Prevention Training and Perineal Massage and Pelvic Floor Exercise
  Interventions: Behavioral: Pelvic Floor Dysfunction Prevention Training; Behavioral: Pelvic Floor Dysfunction Prevention Training and Perineal Massage; Behavioral: Pelvic Floor Dysfunction Prevention Training and Perineal Massage and Pelvic Floor Exercise

INTERVENTIONS:
Behavioral: Pelvic Floor Dysfunction Prevention Training — The "Pelvic Floor Dysfunction Prevention Training" booklet is cover weight control, perineal hygiene, adequate fluid consumption, not smoking and alcohol use, avoidance of spicy, fizzy and fatty foods and beverages, correct posture and frequency of micturition, prevention of constipation and abdominal pressure.
Behavioral: Pelvic Floor Dysfunction Prevention Training and Perineal Massage — Women will apply perineal massage for an average of 8-10 minutes at least twice a week, starting from the 34th week of pregnancy until delivery. In addition to perineal massage, the "Pelvic Floor Dysfunction Prevention Training" booklet will be given to participant.
  Arms: Experimental Group 1; Experimental Group 2
Behavioral: Pelvic Floor Dysfunction Prevention Training and Perineal Massage and Pelvic Floor Exercise — Women assigned to this group will apply pelvic floor exercise at least 3 days a week 8-12 times a week, starting from the 34th week of pregnancy until delivery. In addition, women will apply perineal massage for an average of 8-10 minutes at least twice a week, starting from the 34th week of pregnancy until delivery. In addition to perineal massage, the "Pelvic Floor Dysfunction Prevention Training" booklet will be given to participant.
  Arms: Experimental Group 2

SUMMARY:
This study aimed to determine the effect of perineal massage and pelvic floor exercise in the antenatal period on sexuality and urinary and fecal incontinence in the postpartum period. This study will be conducted in a pregnant school at a state hospital in Turkey. An active control group will be formed as the control group. The control group will be given the "Pelvic Floor Dysfunction Prevention Training" booklet prepared by the researchers. Experimental 1 group will receive perineal massage training in addition to the "Pelvic Floor Dysfunction Prevention Training" booklet given to the control group. Experimental 2 group will receive pelvic floor exercises in addition to perineal massage training and the "Pelvic Floor Dysfunction Prevention Training" booklet given to the control group.

DETAILED DESCRIPTION:
The research was conducted as a randomized controlled trial. The simple randomization method will be used for the assignment to groups. The data of the research; will be collected using the Preliminary Evaluation Form, Personal Information Form, Female Sexual Function Index, The International Consultation on Incontinence Questionnaire-ICIQ-SF (Turkish Version), and Fecal Incontinence Severity Index. The research will start at the 34th week of pregnancy and the questionnaires will be administered in the 3rd month after delivery. There will be 3 groups in the research.An active control group will be formed as the control group. The control group will be given the "Pelvic Floor Dysfunction Prevention Training" booklet prepared by the researchers. Experimental 1 group will receive perineal massage training in addition to the "Pelvic Floor Dysfunction Prevention Training" booklet given to the control group. Experimental 2 group will receive pelvic floor exercises in addition to perineal massage training and the "Pelvic Floor Dysfunction Prevention Training" booklet given to the control group.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old,
* being 32-34th pregnancy weeks,
* being not experiencing any complications in the mother and fetus during pregnancy (gestational diabetes, hypertension, preeclampsia, intrauterine growth retardation, congenital anomaly, etc.),
* having a singleton pregnancy,
* being primiparous
* being volunteer to participate in the study

Exclusion Criteria:

* elective cesarean section planning,
* having a history of chronic constipation,
* having a previous history of urinary or anal incontinence,
* having genital infection with lesions (HSV, HPV, Syphilis, Candida Albicans, Chancroid)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 75 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index | Postpartum 12th weeks
  In the structure of the scale; There are 6 sub-dimensions: desire, arousal, lubrication (lubrication, wetting), orgasm, satisfaction and pain.The highest raw score that can be obtained from the scale is 95 and the lowest raw score is 4.After sub-dimension averages were multiplied by factor loads, the highest score that could be obtained from the scale was calculated as 36 and the lowest score as 2. High score means better function.
The International Consultation on Incontinence Questionnaire-ICIQ | Postpartum 12th weeks
  The International Consultation on Incontinence Questionnaire-ICIQ-SF (Turkish Version) is a scale for evaluating every aspect of urinary incontinence and its impact on quality of life.It consists of 6 questions.The ICIQ Total Score is calculated by the sum of the 3+4+5 questions and scores between 0 and 21. If the score is high and close to 21, it shows that it is overly affected.
Fecal Incontinence Severity Index-FISI | Postpartum 12th weeks
  It is an index developed to diagnose the frequency and type of fecal incontinence.It defines the type of fecal incontinence in four types and its frequency in five categories. The index score is calculated by summing the numbers corresponding to each box and the patient score. In patient-weighted scoring, the highest score that can be obtained from the index is 61 and the lowest score is 0.The cut-off score of the index is 31.7.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Özkan Şat, Dr, Principal Investigator — Bitlis Eren University
Locations (1):
- Karabük Health and Training Hospital, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No